CLINICAL TRIAL: NCT04246749
Title: A Phase 1, Open-label, Two-cohort, Single Dose Study to Assess the Mass Balance, Route of Elimination, and Metabolic Profile of [14C] Labeled CRN00808 and Absolute Bioavailability of CRN00808 in Healthy Male Volunteers
Brief Title: Mass Balance and Pharmacokinetics of [14C]-CRN00808 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Crinetics Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRN00808-06
Record Dates: First submitted 2020-01-14; First posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: [14C]-CRN00808 Oral Solution (Experimental): Single oral dose of CRN00808 containing [14C]-CRN00808
  Interventions: Drug: [14C]-CRN00808
- Part B: CRN00808 Oral Capsule w/ [14C]-CRN00808 IV microtracer (Experimental): Single oral dose of CRN00808 followed by [14C]-CRN00808 IV microtracer injection
  Interventions: Drug: [14C]-CRN00808; Drug: CRN00808

INTERVENTIONS:
Drug: [14C]-CRN00808 — Investigational drug
Drug: CRN00808 — Investigational drug
  Arms: Part B: CRN00808 Oral Capsule w/ [14C]-CRN00808 IV microtracer

SUMMARY:
A phase 1 healthy volunteer study to assess the mass balance, elimination, and metabolic profile of CRN00808. The study will be conducted in 2 parts: Part A, to characterize the absorption, distribution, metabolism, excretion, and mass balance of orally administered radio-labeled CRN00808; Part B, to determine the absolute bioavailability of CRN00808 administered using CRN00808 and radio-labeled CRN00808 as intravenous and oral forms.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects 19 to 55 years of age
2. BMI 18 to 30 kg/m2

Exclusion Criteria:

1. Any uncontrolled or active major systemic disease including, but not limited to: acromegaly (with or without pituitary surgery or radiation therapy), cardiac, pulmonary, gastrointestinal, metabolic, urogenital, neurological, immunological, psychiatric, or neoplastic disorder with metastatic potential
2. History or presence of malignancy within the past 5 years. Subjects who have been successfully treated (for 3 months or longer) with no recurrence of basal or squamous cell carcinoma of the skin or carcinoma in-situ of the cervix may be enrolled.
3. Use of any investigational drug within the past 60 days or 5 half-lives, whichever is longer
4. Have a medically significant abnormality observed during screening or the admission physical examination or in any other baseline measurements
5. Use of any prior medication without approval of the investigator within 14 days prior to admission
6. Tested positive at screening for HIV, hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCV-Ab) or has a history of a positive result
7. History of alcohol or substance abuse in the past 6 months
8. Any condition that in the opinion of the investigator would jeopardize the subject's appropriate participation in this Phase 1 study

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Mass balance of CRN00808 | Up to 21 days (until >90% of dose is recovered)
  Total radioactivity in urine and feces following a single oral dose [14C]-CRN00808 (expressed as a percentage of the total radioactive dose administered)
Absolute bioavailability of CRN00808 | 5 days
  Absolute bioavailability is calculated from the areas under the curve of intravenous and oral administration

SECONDARY OUTCOMES:
Pharmacokinetics (AUC) | Part A: Day 1 to day 21 (depending on recovery of dose). Part B: Day 1 through to Day 7
  Assessment of the plasma area under the curve of CRN00808 and [14C]-CRN00808
Pharmacokinetics (t1/2) | Part A: Day 1 to day 21 (depending on recovery of dose). Part B: Day 1 through to Day 7
  Assessment of the total elimination half-life of CRN00808 and [14C]-CRN00808
Pharmacokinetics (Tmax) | Part A: Day 1 to day 21 (depending on recovery of dose). Part B: Day 1 through to Day 7
  Assessment of Time to attain maximum observed plasma concentration of CRN00808 and [14C]-CRN00808
Pharmacokinetics (CL) | Day 1 through to Day 7
  Assessment of the clearance of CRN00808 (Part B only)
Pharmacokinetics (CL/F) | Part A: Day 1 to day 21 (depending on recovery of dose). Part B: Day 1 through to Day 7
  Assessment of Apparent oral clearance of CRN00808
Pharmacokinetics (Vz) | Day 1 through to Day 7
  Assessment of Volume of distribution at terminal phase (Part B only)
Pharmacokinetics (Vz/F) | Part A: Day 1 to day 21 (depending on recovery of dose). Part B: Day 1 through to Day 7
  Assessment of Apparent volume of distribution at terminal phase

CONTACTS AND LOCATIONS:
Locations (1):
- PRA Health Sciences, Groningen, Netherlands